CLINICAL TRIAL: NCT05232877
Title: Effects of t-DCS Combined With Concurrent Cognitive Training on Apathy in Elderly Subjects With Minor Neurocognitive Impairment
Brief Title: Effects of t-DCS and Cognitive Training on Apathy in Elderly With Minor Neurocognitive Impairment
Acronym: FAME3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-PP-15
Record Dates: First submitted 2021-12-21; First posted 2022-02-10 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Apathy; Neurocognitive Disorders
MeSH Terms: conditions — Lethargy; Neurocognitive Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The intervention group will follow sessions of tDCS combined with a simultaneous cognitive training on tablet.
  he control group will follow cognitive training with a combined sham tDCS. Intervention will last for 4-week with 3 sessions per week (12 sessions).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS combined with simultaneous cognitive training (Experimental)
  Interventions: Other: tDCS
- cognitive training with a combined sham tDCS (Sham Comparator)
  Interventions: Other: SHAM tDCS

INTERVENTIONS:
Other: SHAM tDCS — The control group will follow cognitive training with a combined sham tDCS. Intervention will last for 4-week with 3 sessions per week (12 sessions).
  Arms: cognitive training with a combined sham tDCS
Other: tDCS — The intervention group will follow sessions of tDCS combined with a simultaneous cognitive training on tablet
  Arms: tDCS combined with simultaneous cognitive training

SUMMARY:
Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique using a low intensity electric current to modify cortical excitability. Apathy is a pervasive neuropsychiatric symptom characterized by a reduction in goal-directed behavior and activity that persists over time and causes identifiable functional impairment. The aim of this study is to evaluate the effects of repeated sessions of tDCS combined with simultaneous cognitive training on apathy in older people with minor neurocognitive disorders.

DETAILED DESCRIPTION:
Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation technique using a low intensity electric current to modify cortical excitability. There is growing interest for tDCS for psychiatric illnesses, notably for depression.

Apathy is a pervasive neuropsychiatric symptom characterized by a reduction in goal-directed behavior and activity that persists over time and causes identifiable functional impairment. tDCS could be a promising new area for non-pharmacological treatment of apathy.

The aim of this study is to evaluate the effects of repeated sessions of tDCS combined with simultaneous cognitive training on apathy in older people with minor neurocognitive disorders. For this, 30 apathetic subjects with minor neurocognitive disorders will be included and randomized between two groups. The intervention group will follow sessions of tDCS combined with a simultaneous cognitive training on tablet. The control group will follow cognitive training with a combined sham tDCS. Intervention will last for 4-week with 3 sessions per week (12 sessions). Stimulation will be performed with Startim 20 (Neuroelectrics®) which is approved by the European Union as a Class IIa medical device and meeting European safety standards. Stimulation will last for 20 minutes and the dorsolateral prefrontal cortex (F3) will be targeted. For the intervention group, the electric current will be 2mA. Assessments will be done at baseline, just after the end of intervention and 3 months after intervention. Apathy, daily functional motor behaviors, cognitive functions and fatigue will be assessed with clinician assessment, self-administered questionnaires, ambulatory actigraphy and cognitive tests. The assessments and the intervention will be done by different people. Study will be a double-blind randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Subject consulting in one of the investigating centers
* Clinical diagnosis of Minor Neurocognitive Disorder according to DSM 5 criteria (APA, 2013)
* Apathetic syndrome defined according to the Diagnostic Criteria for Apathy (Miller & al., 2021)
* Subject who can read and write French
* Subjects who are beneficiaries of a social security plan
* Signature of free and informed consent

Exclusion Criteria:

* Current clinical diagnosis of a depressive episode characterized by DSM 5 criteria (APA, 2013)
* Known diagnosis of schizophrenia, bipolar disorder, substance abuse or dependence
* Significant sensory or motor impairment
* Subject under guardianship, conservatorship, or conservatorship
* Active smoking or smoking cessation of less than one year
* Contraindications to the practice of tDCS: history of intracranial hypertension, neurosurgery, metallic implant at the cephalic level, pacemaker
* Unbalanced epilepsy
* Severe somatic disease not stabilized
* Previous use of tDCS (problem of maintaining the integrity of the blinding procedure)
* Scalp skin disease
* Concurrent participation in another drug research study or any other study that may interfere with study results

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-04-05 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2026-06-10 (Estimated)

PRIMARY OUTCOMES:
Apathy Inventory (Robert et al., 2002), clinician version | Changes from baseline severity of apathy at 4 weeks and 18 weeks are assessed (12 weeks after the end of intervention)
  The Apathy Inventory scored from 0 (No problem) to 4 (major problem) the 3 dimensions of apathy: the emotional blunting, the loss of initiative and the loss of interest. A higher total score indicates a greater severity.

SECONDARY OUTCOMES:
Assessment of neuropsychiatric symptoms | Changes from baseline severity of apathy at 4 weeks and 18 weeks are assessed (12 weeks after the end of intervention)
  Clinician assess behavioral symptoms and scored the severity from 0 to 3.
Assessment of the global cognitive functioning | Changes from baseline severity of apathy at 4 weeks and 18 weeks are assessed (12 weeks after the end of intervention)
  Mini mental state examination (MMSE): test for asses the global cognitive functioning
  Unit of measure: score
  Scored from 0 to 30. A lower score indicate lower performance in global cognitive functioning.
Assessment of cognitive functions with FAB | Changes from baseline severity of apathy at 4 weeks and 18 weeks are assessed (12 weeks after the end of intervention)
  Frontal assessment battery (FAB): test for asses global executive functions
  Unit of measure: score
  Scored from 0 to 18. A lower score indicate lower performance in global executive functions.
Assessment of episodic memory | Changes from baseline severity of apathy at 4 weeks and 18 weeks are assessed (12 weeks after the end of intervention)
  Grober and Bruschke test : test for asses episodic memory
  Unit of measure: score
  Scored from 0 to 48. A lower score indicate lower performance in episodic memory
Assessment of attention and mental flexibilty | Changes from baseline severity of apathy at 4 weeks and 18 weeks are assessed (12 weeks after the end of intervention)
  Trail Making test A_b: test for attention and mental flexibilty
  Unit of measure: time to realize the test
  A longer time indicate a lower performance in attention and mental flexibility.
Assessment of working memory | Changes from baseline severity of apathy at 4 weeks and 18 weeks are assessed (12 weeks after the end of intervention)
  Empan de chiffres: test for asses working memory
  Unit of measure: score
  A lower score indicate a lower performance in working memory
Assessment of verbal fluency | Changes from baseline severity of apathy at 4 weeks and 18 weeks are assessed (12 weeks after the end of intervention)
  Fluency test: test for asses verbal fluency
  Unit of measure: number of words produced by the participant into 60 seconds
  A lower score indicate a lower performance.
Assessment of language | Changes from baseline severity of apathy at 4 weeks and 18 weeks are assessed (12 weeks after the end of intervention)
  Test de "dénomination d'image": test for asses language
  Unit of measure: score
  A lower score indicate a lower performance.
Assessment of fatigue with Multidimensional fatigue inventory (MFI) | Changes from baseline severity of apathy at 4 weeks and 18 weeks are assessed (12 weeks after the end of intervention)
  Multidimensional fatigue inventory (MFI): 20-item self-report questionnaire for measuring five dimensions of fatigue.
  Each subscale contains four items, which are scored on a five-point Likert-scale.
  Scores range from 4 (absence of fatigue) to 20 (maximum fatigue) for each subscale.
  Unit of measure: score
Assessment of fatigue with 15-sec Sustained maximal handgrip contraction | Changes from baseline severity of apathy at 4 weeks and 18 weeks are assessed (12 weeks after the end of intervention)
  15-sec Sustained maximal handgrip contraction: The decrease in force during the 15-s was used as the indicator of fatigability.
  Measure: performance for the test: The decrease in force during the 15-s was used as the indicator of fatigability. It was computed as the difference between the area under constant curve equal to the maximal grip force and the area under the force-time curve of 15-s
Assessment of daily physical activity | Changes from baseline severity of apathy at 4 weeks and 18 weeks are assessed (12 weeks after the end of intervention)
  Actigraphy: assessment of time physical activity of light, moderate and vigorous intensity and sedentary time in daily life in minute and % of daily activity.
Assessment of tDCS adverse effects questionnaire | Changes from baseline severity of apathy at 4 weeks and 18 weeks are assessed (12 weeks after the end of intervention)
  tDCS adverse effects questionnaire: questionnaire for asses the tDCS adverse effects.
  It is a 11-item scale. Each item corresponds to an adverse effect. Each item is scored from 1 (absence of the adverse effect) to 4 (severe). If the adverse effect is present (score>1) the clinician scored if this is related to tdCS from 0 (none) to 5 (definite).
  A higher score indicate more adverse effects.
  Unit of measure: score

CONTACTS AND LOCATIONS:
Overall Officials: Eric ETTORE, MD, Principal Investigator — Nice University Hospital
Locations (1):
- Centre Memoire Ressources et Recherche, CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No